CLINICAL TRIAL: NCT05547165
Title: Percutaneous Intervention Versus Observational Trial of Arterial Ductus in Low Weight Infants
Acronym: PIVOTAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Abbott (Industry); University of Pittsburgh (Other); University of Bristol (Other); Dartmouth College (Other); University of Iowa (Other); Emory University (Other); Cedars-Sinai Medical Center (Other); Children's Hospital Los Angeles (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Carl Backes, MD, Professor of Pediatrics, Departments of Neonatology and Cardiology, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00002501; UG3HL161338 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Ductus Arteriosus, Patent
Keywords: PDA
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Primary Comparator (Active Comparator): Interventional groups that subject will be randomly assigned to include Percutaneous Patent Ductus Arteriosus Closure (PPC) or Responsive Management. Those assigned to PPC will undergo active intervention to close a hemodynamically significant patent ductus arteriosus (HSPDA) whereas those assigned to Responsive Management will be treated to manage the symptoms of the HSPDA and permit natural closure over time.
  Interventions: Device: Percutaneous Patent Ductus Arteriosus Closure (PPC); Combination Product: Responsive Management Intervention; Diagnostic Test: Echocardiogram, cardiac
- Secondary Intervention (Other): Sub-group of patients initially randomized to Responsive Management who may suffer a decline in health status that can be attributed to the presence of a hemodynamically significant patent ductus arteriosus (HSPDA). These patients, upon meeting pre-specified clinical criteria, will undergo active treatment via Percutaneous Patent Ductus Arteriosus Closure (PPC) as in the active comparator arm.
  Interventions: Device: Percutaneous Patent Ductus Arteriosus Closure (PPC); Diagnostic Test: Echocardiogram, cardiac

INTERVENTIONS:
Device: Percutaneous Patent Ductus Arteriosus Closure (PPC) — Infants in this group will undergo catheter-based PPC closure ≤48 hours following randomization and within 7-days of qualifying ECHO. All participants assigned to PPC will receive the Amplatzer Piccolo™ Occluder which will be implanted within the duct (intraductal placement). The Piccolo™ occluder is approved by the US FDA for this purpose.
Combination Product: Responsive Management Intervention — Interventional PDA-closure, including PPC or surgical ligation and post-randomization pharmacologic (NSAID or acetaminophen) (enteral or intravenous) PDA treatment, are not allowed unless secondary treatment thresholds (see below) are met. Healthcare decisions for Responsive Management will be made at the discretion of the treatment team, while the infant is carefully monitored for any decline in status that may be attributed to the presence of PDA, in which case, Secondary Intervention (described below) may be considered.
  Despite widespread acceptance of responsive PDA management, no consensus definition exists. The following Responsive Management interventions are permitted but not required per clinician discretion: 1) fluid restriction between 120-140 mL/kg/day; 2) diuretics (per local practice); 3) increases in positive end-expiratory pressure (PEEP).
  Arms: Primary Comparator
Diagnostic Test: Echocardiogram, cardiac — An echocardiogram, also known as "ECHO", is an ultrasound image of the heart. Echocardiography is a common test used for the diagnosis and management of cardiac diseases or conditions.

SUMMARY:
Patent Ductus Arteriosus is a developmental condition commonly observed among preterm infants. It is a condition where the opening between the two major blood vessels leading from the heart fail to close after birth. In the womb, the opening (ductus arteriosus) is the normal part of the circulatory system of the baby, but is expected to close at full term birth. If the opening is tiny, the condition can be self-limiting. If not, medications/surgery are options for treatment.

There are two ways to treat patent ductus arteriosus - one is through closure of the opening with an FDA approved device called PICCOLO, the other is through supportive management (medications). No randomized controlled trials have been done previously to see if one of better than the other. Through our PIVOTAL study, the investigators aim to determine is one is indeed better than the other - if it is found that the percutaneous closure with PICCOLO is better, then it would immediately lead to a new standard of care. If not, then the investigators avoid an invasive costly procedure going forward.

ELIGIBILITY:
Inclusion Criteria:

1. EPIs born between 22-weeks+0 days (220/7 wks) and 27-weeks+6 days (276/7 wks) gestation, inclusive
2. Admitted to a study NICU
3. Birth weight ≥700-grams
4. Mechanically ventilated at time of consent and randomization
5. HSPDA ("PDA Score" ≥6) noted on echocardiogram (ECHO)
6. Randomization is able to be performed within 5 days of the qualifying ECHO and when infant is 7-32 days postnatal

Exclusion Criteria:

Clinical Exclusion Criteria

1. Life-threatening congenital defects (including congenital heart disease such as aortic coarctation or pulmonary artery stenosis). PDA and small atrial/ventricular septal defects are permitted;
2. Congenital lung abnormalities, (e.g. restrictive lung disease);
3. Pharyngeal or airway anomalies (tracheal stenosis, choanal atresia);
4. Treatment for acute abdominal process (e.g., necrotizing enterocolitis);
5. Infants with planned surgery;
6. Active infection requiring treatment;
7. Chromosomal defects (e.g., Trisomy 18);
8. Neuromuscular disorders;
9. Infants whose parents have chosen to allow natural death (do not resuscitate order) or for whom limitation of intensive care treatment is being considered (e.g. severe intraventricular hemorrhage)
10. Physician deems that the infant would not be a Percutaneous PDA Closure candidate due to clinical instability; however, if the infant's clinical status improves before 30-days postnatal and all inclusion criteria are still met, then the infant may be enrolled.

ECHO-based Exclusion Criteria

1. Pulmonary hypertension (defined by ductal right to left shunting for >33% of the cardiac cycle) in which early PDA closure may increase right ventricular afterload and compromise pulmonary and systemic blood flow;
2. Evidence of cardiac thrombus that might interfere with device placement;
3. PDA diameter larger than 4 mm at the narrowest portion (consistent with FDA-approved instructions for Piccolo™ device use).
4. PDA length smaller than 3 mm (consistent with FDA-approved instructions for Piccolo™ device use).
5. PDA that does not meet inclusion requirements ("PDA Score" <6).* * If a potential participant is found to have a PDA meeting eligibility requirements on a subsequent ECHO during the required period of 7 - 30 postnatal days of age, they may then be declared eligible to participate and enrolled, provided all other inclusion criteria are met and exclusion criteria are not met.

Other Exclusion Criteria

1. Parents or legal guardian do not speak English or Spanish

Ages: 7 Days to 32 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of days free of ventilatory support requirement (ventilator-free days; VFDs) | 30 days post-randomization
  Ventilator free days (VFDs) are defined as the number of days that a subject is alive and free from mechanical ventilatory support. VFDs are an established respiratory outcome measure in pediatric clinical trials, and are a strong predictor of short-term and longer-term oucomes, including length of neonatal intensive care unit (NICU) stay, morbidities, and mortality.

SECONDARY OUTCOMES:
Positive-pressure dependency or death | 36 weeks post-menstrual age
  A composite outcome measure (yes/no), positive pressure dependency at 36 weeks post-menstrual age (PMA) is an indicator of chronic lung disease (CLD), the most common and serious respiratory complication of prematurity. Both invasive and non-invasive positive pressure ventilation at 36 weeks PMA is associated with long-term respiratory and neurodevelopmental impairment.
Diagnosis of pulmonary hypertension or death | 36 weeks post-menstrual age
  A compositve binary outcome measure (yes/no), diagnosis of pulmonary hypertension will be determined by cardiac echocardiogram at 36 weeks post-menstrual age. Diagnosis of pulmonary hypertension is an indicator of increased pulmonary vasculature resistance, a marker for increased morbidity and mortality among infants with chronic lung disease.
Total days on mechanical ventilation | 4 months corrected age
  The total number of days (continuous variable) a study subject requires any use of invasive mechanical ventilatory support within a 24-hour calendar day.
Days requiring positive-pressure assisted breathing | Randomization through 4 months corrected age
  The sum of days the study subject requires either invasive or non-invasive positive pressure assisted ventilation within a 24 hour calendar day.
Days on supplemental oxygen | Randomization through 4 months corrected age
  Total number of days the study subject requires supplemental oxygen. The subject may be on either invasive or non-invasive ventilatory support during this time. The subject must be free from supplemental oxygen use for a period of at least 24 hours to interrupt or cease counting.
Time to death | Randomization through 4 months corrected age
  A continuous measure, in days, of the time from a study subject's randomization to expiration, if this occurs.
Diagnosis of cardiac dysfunction | 36 weeks post-menstrual age
  A diagnosis of left-ventricular output by echocardiography (ECHO) at 36 weeks post-menstrual age.
Abnormal cardiac remodeling | 36 weeks post-menstrual age
  Finding of left-ventricular end-diastolic volume (LV EDV) >97% on echocardiography (ECHO) at 36 weeks post-menstrual age.
General Movements Assessment (GMA) | 34 - 36 weeks post-menstrual age
  The General Movements Assessment (GMA) is a standardized video-based neurological exam to evaluate the presence of "fidgety" versus "absent fidgety" and "cramped-synchronized" versus "non cramped-synchronized" movement patterns at 34 - 36 weeks post-menstrual age. It is used to assist in the diagnosis of impaired motor neurodevelopment and cerebral palsy.
Need for rescue intervention | Randomization through 4 months corrected age
  Recording of incidence of need for study subjects randomized to Responsive Management to undergo Percutaneous Patent Ductus Arteriosus Closure (PPC) due to decline in health status.
Hammersmith Neonatal Neurological Examination (HNNE) | 34 - 36 weeks post-menstrual age
  The HNNE is a standardized neurological examination of 34 items to evaluate tone, motor patterns, spontaneous movements, reflexes, visual and auditory attention, and behavior.
Hammersmith Infant Neurological Examination (HINE) | 3 - 4 months of corrected age
  The HINE is similar to the HNNE, used to assess neurological function at 3 - 24 months of age, including cranial nerve function, movements, reflexes, protective reactions and behavior, and age-dependent evaluation of gross and fine-motor function.
Infant/Toddler Sensory Profile (Low Registration Domain) | 3 - 4 months of corrected age
  Caregiver questionnaire responses to determine if their infant appropriately processes and responds to environmental stimuli, versus missing or taking longer to respond ("Low Registration"). There are 13 items with scores of 13 - 65 possible; scores of 42 - 51 are considered "Typical performance".
Infant/Toddler Sensory Profile (Sensation Seeking Domain) | 3 - 4 months of corrected age
  Caregiver questionnaire responses to determine if their infant is hyposensitive, seeking additional sensory stimulation. There are 6 items with scores of 6 - 30 possible; scores of 7 - 15 are considered "Typical performance".
Infant/Toddler Sensory Profile (Sensory Sensitivity Domain) | 3 - 4 months of corrected age
  Caregiver questionnaire responses to determine if their infant responds readily to sensory stimulation, without actively avoiding it. There are 12 items with scores of 12 - 60 possible; scores of 45 - 57 are considered "Typical performance)
Infant/Toddler Sensory Profile (Sensation Avoiding Domain) | 3 - 4 months of corrected age
  Caregiver questionnaire responses to determine if their infant avoids sensory stimulation. There are 5 items with scores of 5 - 25 possible; scores of 19 - 25 are considered "Typical performance".
Infant/Toddler Sensory Profile (Low Threshold Domain) | 3 - 4 months of corrected age
  Caregiver questionnaire responses which are the sum of the Sensory Sensitivity and Sensation Avoiding domains). Summed scores of 15 - 85 are possible; summed scores of 64 - 81 are considered "Typical performance".
Baby Care Questionnaire (BCQ) | 3 - 4 months of corrected age
  The BCQ is another caregiver-based questionnaire for parental perspectives of an infant's feeding and sleeping habits. It is used as an evaluation of a parent's reliance upon structure / routines and attunement (dependence upon infant's cues).
Mother-Infant Bonding Scale (MIBS) | 3 - 4 months of corrected age
  The MIBS is an 8-item questionnaire to evaluate a mother's bondedness towards her infant. Responses are scored from 0 to 3 for each item, with a total possible range of 0 - 24. Lower scores indicate more favorable outcomes for mother-infant bondedness, whereas higher scores indicate the potential for difficulties.
Type and incidence of any adverse event | 3 - 4 months of corrected age
  Reporting of type and frequency of any adverse event that occurs during percutaneous closure procedures, and post-procedurally that may be related to the intervention.
Type and incidence of serious adverse event | 3 - 4 months of corrected age
  Reporting of type and frequency of any serious adverse event (e.g., potentially life-threatening change in status) that occurs during percutaneous closure procedures, and post-procedurally that may be related to the intervention.

OTHER OUTCOMES:
Determine whether neurodevelopment at 3-4 months CA is mediated by improved neurodevelopmental profiles at 34-36 weeks PMA. | 34-36 weeks post-menstrual age and 3 - 4 months corrected age
  Analysis of HNNE / HINE scores to determine if neurodevelopmental evaluation scores conducted at 34 - 36 weeks post-menstrual age mediate outcomes at 3 - 4 months corrected age
Evaluation of effect modifiers on primary and secondary outcomes | Birth to 4 months of corrected age
  Examination of the homogeneity of the effect of HSPDA on the primary and secondary outcomes will be carried out in statistical analyses using stratification variables (e.g., gender, gestational age, etc.) and characteristics not balanced through random assignment, if any such imbalances are found.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - University of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Lucille Packard Children's Hospital at Stanford, Palo Alto, California
  - UC Davis Children's Hospital, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Orlando Health, Orlando, Florida
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota, Masonic Children's Hospital, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Medical Center, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Medical City Children's Dallas, Dallas, Texas
  - UT Southwestern Children's Medical Center of Dallas, Dallas, Texas
  - Texas Children's, Houston, Texas
  - Seattle Children's, Seattle, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benitz WE; Committee on Fetus and Newborn, American Academy of Pediatrics. Patent Ductus Arteriosus in Preterm Infants. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-3730. Epub 2015 Dec 15. PMID 26672023
- [Background] Benitz WE. Patent ductus arteriosus: to treat or not to treat? Arch Dis Child Fetal Neonatal Ed. 2012 Mar;97(2):F80-2. doi: 10.1136/archdischild-2011-300381. Epub 2011 Dec 15. PMID 22174019
- [Background] Liebowitz M, Katheria A, Sauberan J, Singh J, Nelson K, Hassinger DC, Aucott SW, Kaempf J, Kimball A, Fernandez E, Carey WA, Perez J, Serize A, Wickremasinghe A, Dong L, Derrick M, Wolf IS, Heuchan AM, Sankar M, Bulbul A, Clyman RI; PDA-TOLERATE (PDA: TOLEave it alone or Respond And Treat Early) Trial Investigators. Lack of Equipoise in the PDA-TOLERATE Trial: A Comparison of Eligible Infants Enrolled in the Trial and Those Treated Outside the Trial. J Pediatr. 2019 Oct;213:222-226.e2. doi: 10.1016/j.jpeds.2019.05.049. Epub 2019 Jun 27. PMID 31255386
- [Background] Donovan JL, Rooshenas L, Jepson M, Elliott D, Wade J, Avery K, Mills N, Wilson C, Paramasivan S, Blazeby JM. Optimising recruitment and informed consent in randomised controlled trials: the development and implementation of the Quintet Recruitment Intervention (QRI). Trials. 2016 Jun 8;17(1):283. doi: 10.1186/s13063-016-1391-4. PMID 27278130
- [Background] Wilson C, Rooshenas L, Paramasivan S, Elliott D, Jepson M, Strong S, Birtle A, Beard DJ, Halliday A, Hamdy FC, Lewis R, Metcalfe C, Rogers CA, Stein RC, Blazeby JM, Donovan JL. Development of a framework to improve the process of recruitment to randomised controlled trials (RCTs): the SEAR (Screened, Eligible, Approached, Randomised) framework. Trials. 2018 Jan 19;19(1):50. doi: 10.1186/s13063-017-2413-6. PMID 29351790
- [Background] Donovan JL, Lane JA, Peters TJ, Brindle L, Salter E, Gillatt D, Powell P, Bollina P, Neal DE, Hamdy FC; ProtecT Study Group. Development of a complex intervention improved randomization and informed consent in a randomized controlled trial. J Clin Epidemiol. 2009 Jan;62(1):29-36. doi: 10.1016/j.jclinepi.2008.02.010. Epub 2008 Jul 10. PMID 18619811
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Background] Rooshenas L, Scott LJ, Blazeby JM, Rogers CA, Tilling KM, Husbands S, Conefrey C, Mills N, Stein RC, Metcalfe C, Carr AJ, Beard DJ, Davis T, Paramasivan S, Jepson M, Avery K, Elliott D, Wilson C, Donovan JL; By-Band-Sleeve study group; CSAW study group; HAND-1 study group; Optima prelim study group; Romio feasibility study group. The QuinteT Recruitment Intervention supported five randomized trials to recruit to target: a mixed-methods evaluation. J Clin Epidemiol. 2019 Feb;106:108-120. doi: 10.1016/j.jclinepi.2018.10.004. Epub 2018 Oct 16. PMID 30339938
- [Background] Donovan JL, Paramasivan S, de Salis I, Toerien M. Clear obstacles and hidden challenges: understanding recruiter perspectives in six pragmatic randomised controlled trials. Trials. 2014 Jan 6;15:5. doi: 10.1186/1745-6215-15-5. PMID 24393291
- [Background] Rooshenas L, Elliott D, Wade J, Jepson M, Paramasivan S, Strong S, Wilson C, Beard D, Blazeby JM, Birtle A, Halliday A, Rogers CA, Stein R, Donovan JL; ACST-2 study group; By-Band-Sleeve study group; Chemorad study group; CSAW study group; Optima prelim study group; POUT study group. Conveying Equipoise during Recruitment for Clinical Trials: Qualitative Synthesis of Clinicians' Practices across Six Randomised Controlled Trials. PLoS Med. 2016 Oct 18;13(10):e1002147. doi: 10.1371/journal.pmed.1002147. eCollection 2016 Oct. PMID 27755555
- [Background] Mills N, Donovan JL, Wade J, Hamdy FC, Neal DE, Lane JA. Exploring treatment preferences facilitated recruitment to randomized controlled trials. J Clin Epidemiol. 2011 Oct;64(10):1127-36. doi: 10.1016/j.jclinepi.2010.12.017. Epub 2011 Apr 7. PMID 21477994
- [Background] Jepson M, Elliott D, Conefrey C, Wade J, Rooshenas L, Wilson C, Beard D, Blazeby JM, Birtle A, Halliday A, Stein R, Donovan JL; CSAW study group; Chemorad study group; POUT study group; ACST-2 study group; OPTIMA prelim study group. An observational study showed that explaining randomization using gambling-related metaphors and computer-agency descriptions impeded randomized clinical trial recruitment. J Clin Epidemiol. 2018 Jul;99:75-83. doi: 10.1016/j.jclinepi.2018.02.018. Epub 2018 Mar 2. PMID 29505860
- [Background] Donovan JL, de Salis I, Toerien M, Paramasivan S, Hamdy FC, Blazeby JM. The intellectual challenges and emotional consequences of equipoise contributed to the fragility of recruitment in six randomized controlled trials. J Clin Epidemiol. 2014 Aug;67(8):912-20. doi: 10.1016/j.jclinepi.2014.03.010. Epub 2014 May 5. PMID 24811157
- [Background] Rooshenas L, Paramasivan S, Jepson M, Donovan JL. Intensive Triangulation of Qualitative Research and Quantitative Data to Improve Recruitment to Randomized Trials: The QuinteT Approach. Qual Health Res. 2019 Apr;29(5):672-679. doi: 10.1177/1049732319828693. Epub 2019 Feb 22. PMID 30791819
- [Background] Coyne IT. Sampling in qualitative research. Purposeful and theoretical sampling; merging or clear boundaries? J Adv Nurs. 1997 Sep;26(3):623-30. doi: 10.1046/j.1365-2648.1997.t01-25-00999.x. PMID 9378886
- [Background] Glaser BG, Strauss AL. The Discovery of Grounded Theory: Strategies for Qualitative Research. Vol. ed.: Aldine; 1967.
- [Background] US Food and Drug Administration. Use of electronic informed consent, questions and answers: Guidance for institutional review boards, investigators, and sponsors. Silver Spring, MD: US Food and Drug Administration. 2016.
- [Background] Lawrence CE, Dunkel L, McEver M, Israel T, Taylor R, Chiriboga G, Goins KV, Rahn EJ, Mudano AS, Roberson ED, Chambless C, Wadley VG, Danila MI, Fischer MA, Joosten Y, Saag KG, Allison JJ, Lemon SC, Harris PA. A REDCap-based model for electronic consent (eConsent): Moving toward a more personalized consent. J Clin Transl Sci. 2020 Apr 3;4(4):345-353. doi: 10.1017/cts.2020.30. PMID 33244416
- [Background] Paramasivan S, Strong S, Wilson C, Campbell B, Blazeby JM, Donovan JL. A simple technique to identify key recruitment issues in randomised controlled trials: Q-QAT - Quanti-Qualitative Appointment Timing. Trials. 2015 Mar 11;16:88. doi: 10.1186/s13063-015-0617-1. PMID 25873096
- [Background] Watterberg KL, Walsh MC, Li L, Chawla S, D'Angio CT, Goldberg RN, Hintz SR, Laughon MM, Yoder BA, Kennedy KA, McDavid GE, Backstrom-Lacy C, Das A, Crawford MM, Keszler M, Sokol GM, Poindexter BB, Ambalavanan N, Hibbs AM, Truog WE, Schmidt B, Wyckoff MH, Khan AM, Garg M, Chess PR, Reynolds AM, Moallem M, Bell EF, Meyer LR, Patel RM, Van Meurs KP, Cotten CM, McGowan EC, Hines AC, Merhar S, Peralta-Carcelen M, Wilson-Costello DE, Kilbride HW, DeMauro SB, Heyne RJ, Mosquera RA, Natarajan G, Purdy IB, Lowe JR, Maitre NL, Harmon HM, Hogden LA, Adams-Chapman I, Winter S, Malcolm WF, Higgins RD; Eunice Kennedy Shriver NICHD Neonatal Research Network. Hydrocortisone to Improve Survival without Bronchopulmonary Dysplasia. N Engl J Med. 2022 Mar 24;386(12):1121-1131. doi: 10.1056/NEJMoa2114897. PMID 35320643
- [Background] Gordon Lan KK, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika. 1983;70(3):659-663.
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] L Orton J, McGinley JL, Fox LM, Spittle AJ. Challenges of neurodevelopmental follow-up for extremely preterm infants at two years. Early Hum Dev. 2015 Dec;91(12):689-94. doi: 10.1016/j.earlhumdev.2015.09.012. Epub 2015 Oct 27. PMID 26513630
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Wasserstein RL, Schirm AL, Lazar NA. Moving to a world beyond "p< 0.05". In. Vol 73: Taylor & Francis; 2019:1-19.
- [Background] Szklo M, Nieto FJ. Epidemiology: Beyond the Basics. Vol. 3rd ed. Burlington, MA: Jones & Bartlett Learning; 2014.
- [Background] Jensen EA, DeMauro SB, Kornhauser M, Aghai ZH, Greenspan JS, Dysart KC. Effects of Multiple Ventilation Courses and Duration of Mechanical Ventilation on Respiratory Outcomes in Extremely Low-Birth-Weight Infants. JAMA Pediatr. 2015 Nov;169(11):1011-7. doi: 10.1001/jamapediatrics.2015.2401. PMID 26414549
- [Background] Vliegenthart RJS, van Kaam AH, Aarnoudse-Moens CSH, van Wassenaer AG, Onland W. Duration of mechanical ventilation and neurodevelopment in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2019 Nov;104(6):F631-F635. doi: 10.1136/archdischild-2018-315993. Epub 2019 Mar 20. PMID 30894396